CLINICAL TRIAL: NCT02519114
Title: Natural Killer Cel Alloreactive Bone Marrow Transplantation for Multiple Myeloma
Brief Title: Haploidentical Bone Marrow Stem Cell Transplantation in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Gerard Bos, Prof Dr, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL49476.000
Record Dates: First submitted 2015-05-28; First posted 2015-08-10 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: M Myeloma; KIR ligand mismatch; Haploidentical
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone MarrowTransplantation (Experimental): KIR-mismatched haploidentical bone marrow transplantation
  Interventions: Procedure: Donor Bone Marrow stem cell transplantation

INTERVENTIONS:
Procedure: Donor Bone Marrow stem cell transplantation — KIR-mismatched haploidentical Bone Marrow stem cell transplantation

SUMMARY:
The aim of this phase 2 study is to demonstrate that KIR-ligand mismatched haploBMT with post-transplant cyclophosphamide will improve progression free survival in poor risk multiple myeloma patients.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effectiveness of a new treatment modality, the KIR-ligand mismatched haploidentical stem cell transplantation (haploBMT), for poor risk multiple myeloma (MM) patients. MM is a malignancy of plasma cells that usually resides in the bone marrow. Despite new treatment modalities that have been introduced in the last years, MM is still an incurable disease for most patients and median survival for the younger patients (<65) is about 5 years. MM can be treated by several disease modifiers - classical chemotherapy, high dose chemotherapy and autologous stem cell transplantation (ASCT), immunomodulators like thalidomide and lenalidomide, and drugs like bortezomib that interact with relevant intracellular pathways of malignant plasma cells. Though these treatment modalities have improved overall survival and quality of life, patients are not cured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MM <60 years.
* Poor prognosis MM patients, permissive for KIR-ligand mismatch and with a KIR-ligand mismatched haploidentical donor. Poor prognosis is based on:

  * Patients with early disease recurrence (within 12 months after first ASCT) or
  * Patients after a minimum of three lines of chemotherapy (including high dose therapy followed by ASCT rescue therapy) or
  * Poor risk based on the cytogenetic profile.
* Written informed consent
* No HLA identical related or 10/10 matched unrelated donor
* Permissive for KIR-ligand mismatch
* Responsive after reinduction therapy
* Measurable disease

Exclusion Criteria:

* - Patients with an full matched (10/10) donor, who will enroll in the HOVON 96 study
* Active uncontrolled infections
* Uncontrolled CNS involvement by the malignant disease
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease)
* Severe pulmonary dysfunction (CTCAE grade III-IV)
* Severe neurological or psychiatric disease
* Significant hepatic dysfunction (serum bilirubin or transaminases ≥ 3 times upper limit of normal)
* Significant renal dysfunction (creatinine clearance < 30 ml/min after rehydration)
* History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma
* Any psychological, familial, lingual, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Breast-feeding female patients.
* Concurrent severe and/or uncontrolled medical condition (DM, hypertension, cancer).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (scale) | 1 year

SECONDARY OUTCOMES:
Response rate (scale) | analyzed at -7, 30, 60, 90, 120, 150, 180, 270 and 360 days post-transplatation
Incidence of graft failure, engraftment and time to neutrophil and platelet recovery (hematology) | 30 days after transplantation
Incidence and Severity of Acute and Chronic GVHD (scale) | analyzed during follow-up of 1,5 years
Non-Relapse Mortality (number) | 1.5 years
Evaluation of infections after haploBMT and T cell reconstitution (scale) | 1 year after transplantation
NK cell repertoire reconstitution and maturation rates including alloreactivity (facs) | 1 year after transplantation
NK cell repertoire in the Bone Marrow before and after transplantation (facs) | 6 weeks after transplantation
Cost calculation (euro) | 1.5 years
Quality of Life (questionnaire) | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Geesing, Study Director — Maastricht Medical University
Locations (1):
- Maastricht university Medical center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Elssen C, van Gorkom G, Voorter C, von dem Borne P, Meijer E, Wieten L, Bos G. Haploidentical transplantation in patients with multiple myeloma making use of natural killer cell alloreactive donors. Ann Hematol. 2021 Jan;100(1):181-187. doi: 10.1007/s00277-020-04303-z. Epub 2020 Oct 28. PMID 33112968